CLINICAL TRIAL: NCT00004853
Title: A Randomized Trial of Filgrastim-SD/01 vs. Filgrastim in Newly Diagnosed Children and Young Adults With Sarcoma Treated With Dose-Intensive Chemotherapy
Brief Title: Comparison of Filgrastim and Filgrastim SD/01in Boosting White Cell Counts After Intensive Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000092; 00-C-0092; NCT00020137 (obsolete NCT alias)
Record Dates: First submitted 2000-03-04; First posted 2000-03-06 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2016-01-27

CONDITIONS: Ewing's Sarcoma; Rhabdomyosarcoma; MPNST; Synovial Sarcoma; High-risk Sarcoma
Keywords: AMGEN; Granulocyte Colony-Stimulating Factor; MPNST; Randomized; Sarcoma; Tumor
MeSH Terms: conditions — Sarcoma, Ewing; Rhabdomyosarcoma; Neurofibrosarcoma; Sarcoma, Synovial; Sarcoma; Neoplasms | interventions — Filgrastim; pegfilgrastim

ARMS (2):
- 1 (Experimental): single dose of intervention after each cycle of Standard 5 drug dose-intensive chemotherapy
  Interventions: Biological: Filgrastim
- 2 (Experimental): single dose of interventionafter each cycle of Standard 5 drug dose-intensive chemotherapy
  Interventions: Biological: Filgrastim-SD/01

INTERVENTIONS:
Biological: Filgrastim — 5 microgram/kg/dose SC daily starting 24-36 hours after last dose of chemotherapy until post-nadir ANC >=10,000/microliter
  Arms: 1
Biological: Filgrastim-SD/01 — 100 microgram/kg SC 24-36 hours after last dose of chemotherapy (single dose)
  Arms: 2

SUMMARY:
Filgrastim (granulocyte colony-stimulating factor), which is administered by daily subcutaneous injection after cytotoxic chemotherapy, shortens the duration of chemotherapy-induced neutropenia and lowers the risk of infection. In children treated with dose-intensive chemotherapy, filgrastim reduces the duration of severe neutropenia and, as a result, has become a standard component of the treatment regimen. Filgrastim-SD/01 (AMGEN), which is produced by PEGylation of the amino-terminus of filgrastim, is a sustained duration form of granulocyte colony-stimulating factor. In phase I and phase II trials in adults, a single dose of Filgrastim-SD/01 appears to be equivalent to daily dosing of filgrastim in enhancing neutrophil recovery and has a comparable adverse event profile.

Dose-intensive vincristine/cyclophosphamide/doxorubicin (VDoxC) alternating with ifosfamide/etoposide (IE) has become standard therapy for children and adolescents with Ewing's sarcoma and other sarcomas treated at the POB/NCI and other cancer centers within the US. Supportive care measures used in children who are treated with this regimen include mesna to prevent oxazaphosphorine urotoxicity, dexrazoxane to reduce doxorubicin cardiotoxicity, and filgrastim to shorten the duration of neutropenia. The purpose of this randomized open label trial is to compare the tolerance, toxicity, and therapeutic effects of Filgrastim-SD/01 given as a single injection after chemotherapy to daily subcutaneous filgrastim in patients with newly diagnosed sarcoma. The pharmacokinetics of Filgrastim-SD/01 will also be compared to the pharmacokinetics of filgrastim. This trial will also be a platform for performing biological studies of these tumors and for detailed cardiac studies. High-risk patients who are treated on this front line trial and respond will also be candidates for a planned transplant protocol. A total of 34 patients (17 patients per treatment arm) will be entered onto the trial.

DETAILED DESCRIPTION:
Background:

* Filgrastim (granulocyte colony-stimulating factor), which is administered by daily subcutaneous injection after cytotoxic chemotherapy, shortens the duration of chemotherapy-induced neutropenia and lowers the risk of infection.
* In children treated with dose-intensive chemotherapy, Filgrastim reduces the duration of severe neutropenia and, as a result, has become a standard component of the treatment regimen.
* Filgrastim-SD/01 (AMGEN), which is produced by PEGylation of the amino-terminus of Filgrastim, is a sustained duration form of granulocyte colony-stimulating factor.
* In phase I and phase II trials in adults, a single dose of Filgrastim-SD/01 appears to be equivalent to daily dosing of Filgrastim in enhancing neutrophil recovery and has a comparable adverse event profile.
* Dose-intensive vincristine/cyclophosphamide/doxorubicin (VDoxC) alternating with ifosfamide/etoposide (IE) has become standard therapy for children and adolescents with Ewing's sarcoma and other sarcomas treated at the POB/NCI and other cancer centers within the US.

Objectives:

* Compare the tolerance, toxicity, and therapeutic effects of Filgrastim-SD/01 given as a single injection after chemotherapy to daily subcutaneous Filgrastim in patients with newly diagnosed sarcoma receiving multi-agent, dose intensive chemotherapy.
* The pharmacokinetics of Filgrastim-SD/01 will also be compared to the pharmacokinetics of Filgrastim.
* This trial will also be a platform for performing biological studies of these tumors study neutrophil function and CD34 mobilization, and for detailed cardiac studies.

Eligibility:

* Children and young adults (less than or equal to 25 years) with previously untreated high-risk sarcomas (Ewing sarcoma, rhabdomyosarcoma, MPNST, and synovial sarcoma).
* No evidence of tumor infiltration of the bone marrow.

Design:

* Participants will be randomized (1:1) to receive a single dose of Filgrastim-SD/01 or daily filgrastim as a SQ injection after each cycle of chemotherapy.
* Standard 5 drug dose-intensive chemotherapy with vincristine, doxorubicin, cyclophosphamide alternating with ifosfamide and etoposide will be administered.
* Surgery or radiation for the primary tumor will occur after cycle 5.
* A total of 34 patients (17 patients per treatment arm) will be entered onto the trial.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Newly diagnosed histologically proven:

  * Ewing's sarcoma family of tumors, including peripheral neuroectodermal tumors;
  * Alveolar rhabdomyosarcoma;
  * Stage 3 or 4 embryonal rhabdomyosarcoma;
  * Malignant peripheral nerve sheath tumor that is unresectable, incompletely resected with bulk residual disease or metastatic;
  * Synovial cell sarcoma that is unresectable, incompletely resected with bulk residual disease, or metastatic.
* Age equal to or less than 25 years at the time of diagnosis.
* Normal cardiac function (ejection fraction by MUGA or ECHO that is within the institutional normal range).
* Normal serum creatinine for age or creatinine clearance greater than 60 ml/min/1.73m(2).
* Normal liver function (SGPT less than 5 times the upper limit of normal and bilirubin less than 2.5 times the upper limit of normal).
* Normal hematologic function (absolute neutrophil count equal to or greater than 1500/microL, hemoglobin equal to or greater than 9.0 g/dl and platelet count equal to or greater than 100,000/microL).
* Subjects of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study.

EXCLUSION CRITERIA:

* Previous chemotherapy or radiotherapy.
* Pregnant or breast feeding females because the chemotherapy administered on this trial could have a detrimental effect on the developing fetus or newborn.
* Histological evidence of tumor infiltration of bone marrow.
* Stage 1 or 2 embryonal rhabdomyosarcomas.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2000-03-03; Primary Completion 2009-05-20 (Actual); Study Completion 2009-05-20 (Actual)

PRIMARY OUTCOMES:
Tolerance and toxicity | 1 year
PKs | 1 year

SECONDARY OUTCOMES:
Compare neutrophil function
Compare CD34 positive stem cell mobilization
Compare days of febrile neutropenia, days on antibiotics, and inpatient days resulting from neutropenia
Evaluate the role of functional cardiac MRI and serum troponin T levels in detecting early doxorubicin cardiotoxicity
Assess methods of detecting minimal residual disease
cDNA microarray analysis of gene expression, development of cell lines and xenotransplantation models, and exploration of apoptotic pathways

CONTACTS AND LOCATIONS:
Overall Officials: Crystal L Mackall, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Delgado C, Francis GE, Fisher D. The uses and properties of PEG-linked proteins. Crit Rev Ther Drug Carrier Syst. 1992;9(3-4):249-304. PMID 1458545
- [Background] Welte K, Gabrilove J, Bronchud MH, Platzer E, Morstyn G. Filgrastim (r-metHuG-CSF): the first 10 years. Blood. 1996 Sep 15;88(6):1907-29. No abstract available. PMID 8822908
- [Background] Layton JE, Hockman H, Sheridan WP, Morstyn G. Evidence for a novel in vivo control mechanism of granulopoiesis: mature cell-related control of a regulatory growth factor. Blood. 1989 Sep;74(4):1303-7. PMID 2475185